CLINICAL TRIAL: NCT05885412
Title: A Phase 1 Dose Escalation Trial Evaluating an Intravenously Administered Recombinant Adeno-Associated Virus Serotype rh.74 (AAVrh.74) Vector Containing the Human Plakophilin-2a (PKP2a) Coding Sequence (RP-A601; AAVrh.74-PKP2a) in Subjects With Arrhythmogenic Cardiomyopathy Arising From Pathogenic PKP2 Variants (PKP2-ACM)
Brief Title: A Phase 1, Dose Escalation Trial of RP-A601 in Subjects With PKP2 Variant-Mediated Arrhythmogenic Cardiomyopathy (PKP2-ACM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP-A601-0323
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: PKP2 Arrhythmogenic Cardiomyopathy (PKP2-ACM)
Keywords: Arrhythmogenic cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy; Arrhythmogenic Right Ventricular Dysplasia; Sudden Cardiac Death; Genetic cardiomyopathy; Gene therapy; PKP2; ARVC; ARVD; ACM; Cardiac Arrest; Ventricular Arrhythmia
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-A601 (Experimental): Single ascending dose of RP-A601 in 2 consecutive cohorts
  Interventions: Genetic: RP-A601

INTERVENTIONS:
Genetic: RP-A601 — RP-A601 is a recombinant viral vector composed of an AAV serotype rh.74 (AAVrh.74) capsid encapsulating the transgene, human plakophilin 2 (PKP2), transcript variant 2a (PKP2a)

SUMMARY:
This Phase 1 dose escalation trial will assess the safety and preliminary efficacy of a single dose intravenous infusion of RP-A601 in high-risk adult patients with PKP2-ACM.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female ≥18 years at the time of signing the informed consent
2. Capable and willing to provide signed informed consent
3. Clinical diagnosis of ACM as defined by the 2010 revised Task Force Criteria (TFC)
4. Documentation of a pathogenic or likely pathogenic truncating variant in PKP2
5. History of Implantable Cardioverter-Defibrillator (ICD) implantation ≥6 months prior to enrollment
6. PVC frequency ≥500 per 24 hours by ambulatory rhythm monitoring
7. Left ventricular ejection fraction by echocardiogram or CMR ≥50%

Key Exclusion Criteria:

1. Anti-AAVrh.74 capsid neutralizing antibody titer of >1:40
2. Cardiomyopathy related to a genetic etiology other than PKP2 truncating variant
3. Previous participation in a study of gene transfer or gene editing
4. Severe Right ventricular (RV) dysfunction
5. New York Heart Association (NYHA) Class IV heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety associated with RP-A601 | 12 months post-infusion
  Incidence of treatment emergent adverse events (TEAEs), incidence of Serious Adverse Events (SAEs), and identification of Dose Limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
Preliminary efficacy of RP-A601 - Myocardial PKP2 protein expression | 12 months post-infusion
  Assessment of changes in myocardial PKP2 protein expression
Preliminary efficacy of RP-A601 - Ventricular ectopy and arrhythmia | 12 months post-infusion
  Assessment of changes in levels of ventricular ectopy and arrhythmia on cardiac rhythm monitoring
Preliminary efficacy of RP-A601 - Cardiac biomarkers | 12 months post-infusion
  Assessment of changes in circulating levels of cardiac biomarkers of injury and stress

CONTACTS AND LOCATIONS:
Overall Officials: Barry Greenberg, MD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - Duke University, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania